CLINICAL TRIAL: NCT02744989
Title: STIM'ZO : Examining tDCS as an add-on Treatment for Persistent Symptoms in Schizophrenia (SCH)
Brief Title: STIM'ZO : Examining tDCS as an add-on Treatment for Persistent Symptoms in Schizophrenia
Acronym: STIM'ZO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 69HCL14_0446
Record Dates: First submitted 2016-03-18; First posted 2016-04-20 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Mental Disorders; Schizophrenia
Keywords: Schizophrenia; Transcranial direct-current stimulation (tDCS); Sham; Positive and Negative Syndrome Scale (PANSS); Functional Magnetic Resonance Imaging (fRMI); Brain-Derived-Neurotrophic Factor (BDNF)
MeSH Terms: conditions — Mental Disorders; Schizophrenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active tDCS (Experimental): Stimulation will be performed using an tDCS stimulator (Neuroconn or Neuroelectric tDCS stimulator) with two 7×5 cm (35 cm2) sponge electrodes soaked in a saline solution (0.9% NaCl). The anode will be placed with the middle of the electrode over a point midway between F3 and FP1 (left prefrontal cortex: dorsolateral prefrontal cortex, assumed to correspond to a region including Brodmann's Areas (BA) 8, 9, 10, and 46, depending on the patient). The cathode will be located over a point midway between T3 and P3 (left temporo-parietal junction, assumed to correspond to a region including BA 22, 39, 40, 41, and 42, depending on the patient). The stimulation level will be set at 2 mA for 20 minutes during stimulation sessions twice a day for 5 consecutive weekdays. The twice daily sessions will be separated by at least 2 hours.
  Interventions: Device: Neuroconn or Neuroelectric tDCS stimulator
- Sham tDCS (Sham Comparator)
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Neuroconn or Neuroelectric tDCS stimulator — Stimulation parameters were chosen in conformity with those for the treatment of schizophrenic symptoms (Brunelin et al, 2012), adapted according to the latest data from the literature and the tDCS operating stimulator. The experimental tDCS group will receive the ACTIVE stimulation with the following parameters: oscillatory Direct Current with high frequency random noise stimulation (hf-tRNS - 100 to 500 Hz), Intensity = 2 mA, offset = + 1 mA, seance duration = 20 minutes ramp up/ramp down 30 seconds. Total number of sessions = 10 (sessions twice daily for 5 days separated by at least 2 hours for 5 consecutive weekdays).
  Arms: Active tDCS
Device: Sham tDCS — The control group will receive the SHAM stimulation (placebo) following the same regimen (i.e., twice daily sessions separated by at least 2 hours for 5 consecutive weekdays). Sham stimulation consists of a 20 minutes session including 40 seconds of active stimulation (same parameters as in the ACTIVE arm) at the beginning of the sessions, whatever the stimulator
  Arms: Sham tDCS

SUMMARY:
This project aims to provide the proof of concept for transcranial direct-current stimulation (tDCS) in the treatment of resistant/persistent Schizophrenia symptoms. The purpose is to investigate the effect of tDCS on symptoms in schizophrenic patients demonstrating a partial response to a first frequently prescribed antipsychotic medication. An early optimization of the therapeutic strategy must constitute an important factor for prognosis. Hypothesize is that tDCS should alleviate symptoms in patients depending on the clinical characteristics. In this study, stimulation is an add-on treatment to antipsychotic medication, and will be used in a broad variety of patients, i.e. in patients with varied durations of illness, various symptoms profiles, and various levels of treatment response. This in turn will allow the determination of the extent to which results can be generalized to varied patient populations, as well as the extent to which various therapeutic targets (e.g. different symptom dimensions, cognitive performance and brain connectivity) may be improved with tDCS. Despite interesting preliminary results, our team is unable to describe optimal non-invasive brain stimulation (NIBS) response markers.

This study is a randomized, double blind, controlled, French multicenter study (11 centers). The investigators plan to include 144 patients with persistent symptoms in schizophrenia. Seventy two subjects will receive active tDCS and 72 subjects will receive sham tDCS (placebo). Hypothesize is a lasting effect of active tDCS on the schizophrenic symptoms as measured by the number of responders, defined as a decrease of at least 25% of symptoms as measured by a standardized clinical scale score (PANSS) between baseline and after the 10-session tDCS regimen.

Furthermore, the participants believe that an in depth understanding of the cortical effects of tDCS could constitute an important step towards improving the technique and developing treatment response markers. An analysis of the effects on cortical activity and plasticity markers could be an interesting approach.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of schizophrenia according to DSM 5.0 (Diagnostic and Statistical Manuel 5.0) criteria
2. Presence of symptoms despite the optimization of the antipsychotic dosage (based on prescriber's judgment) for at least 6 weeks, i.e. a dosage increase cannot be considered due to tolerability issues and/or is judged unlikely to bring sufficient clinical improvement. This will be operationalized by a minimum Negative PANSS score of 20 and at least one item scoring > 4; OR a minimum Positive PANSS score of 20 with at least one item scoring > 4 (e.g. delusion or hallucination), indicating persistent negative symptoms and/or persistent positive symptoms,
3. Patient under curatorship/guardianship or not
4. Age between 18 and 65 years old.
5. Covered by, or having the right to Social Security
6. Patient who understands the French language
7. Informed consent signed

Exclusion Criteria:

1. Other neuropsychiatric disorders (psychiatric history will be assessed using the MINI 6.0 (Mini International Neuropsychiatric Interview 6.0)) including bipolar disorders and mood depression disorders - (NB: Patients with substance related and addictive disorders will not be excluded from the study, but these data will be carefully recorded).
2. Contraindications for tDCS (neurologic stimulator, pacemaker, cardiac defibrillator, cardiac prosthesis, vascular prosthesis, intracranial clips or clamps, cerebrospinal fluid derivation, metallic splinters in the eyes),
3. Increase in total composite PANSS score of at least 20% between screening and enrollment visits
4. Women who are pregnant
5. Patients whose clinical condition requires in patient procedure under constraint

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2022-05 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Number of responders | Between baseline (day 0) and after 10-sessions of tDCS regimen (day 5)
  The number of responders is based on the Positive and Negative Syndrome Scale (PANSS) score in the active and the sham group after 5 days of tDCS.
  According to Leucht et al (2009), response is defined as a decrease of at least 25% in the Positive and Negative Syndrome Scale (PANSS, Kay et al., 1987) score after the intervention.

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) score | Baseline, day 5 (after 10-sessions of tDCS regimen), 1 month, 3 months and 6 months after the last tDCS session
  Long-term clinical efficacy of active tDCS on schizophrenic symptoms is assessed by PANSS score measured between baseline (day 0), after 10-sessions of tDCS regimen (day 5), 1 month after tDCS (day 30), 3 months after tDCS (day 90) and 6 months after tDCS (day 180).
  The PANSS is a 30-item rater-administered assessment scale of the psychopathological symptoms observed in patients experiencing psychotic states, in particular schizophrenia. The items are noted from 1 to 7. It allows the calculation of the scores for three syndromic dimensions (positive, negative, and general psychopathology), both from a categorical and dimensional perspective. It is particularly recommended for determining a psychopathological profile, to look for predictive elements of an evolution, and to evaluate the respective efficacies of diverse therapeutic strategies.
Auditory Hallucination Rating Scale (AHRS) score | Baseline, day 5 (after 10-sessions of tDCS regimen), 1 month, 3 months and 6 months after the last tDCS session
  Long-term clinical efficacy of active tDCS on schizophrenic symptoms is assessed by AHRS score measured between baseline (day 0), after 10-sessions of tDCS regimen (day 5), 1 month after tDCS (day 30), 3 months after tDCS (day 90) and 6 months after tDCS (day 180).
  The AHRS score measures the severity of auditory hallucinations.
Psycho-Sensory hAllucinations Scale (PSAS) score | Baseline, day 5 (after 10-sessions of tDCS regimen), 1 month, 3 months and 6 months after the last tDCS session
  Long-term clinical efficacy of active tDCS on schizophrenic symptoms is assessed by PSAS score measured between baseline (day 0), after 10-sessions of tDCS regimen (day 5), 1 month after tDCS (day 30), 3 months after tDCS (day 90) and 6 months after tDCS (day 180).
  The PSAS score measures the delusions and severity of hallucinations
Calgary Depression Scale for Schizophrenia (CDSS) score | Baseline, day 5 (after 10-sessions of tDCS regimen), 1 month, 3 months and 6 months after the last tDCS session
  Long-term clinical efficacy of active tDCS on schizophrenic symptoms is assessed by CDSS score measured between baseline (day 0), after 10-sessions of tDCS regimen (day 5), 1 month after tDCS (day 30), 3 months after tDCS (day 90) and 6 months after tDCS (day 180).
  The CDSS score measures depression.
Clinical Global Impression (CGI) score | Baseline, day 5 (after 10-sessions of tDCS regimen), 1 month, 3 months and 6 months after the last tDCS session
  Long-term clinical efficacy of active tDCS on schizophrenic symptoms is assessed by CGI score measured between baseline (day 0), after 10-sessions of tDCS regimen (day 5), 1 month after tDCS (day 30), 3 months after tDCS (day 90) and 6 months after tDCS (day 180).
  The CGI score measures the severity of symptoms and response to treatment.
Shortened Quality of Life questionnaire score | Baseline and 6 months after the last tDCS session
  Quality of life is assessed by S-QoL18 (Shortened Quality of Life questionnaire) scale. S-QoL18 scale assesses eight dimensions : psychological well-being, self-esteem, family relationships, relationships with friends, resilience, physical well-being, autonomy and sentimental life.
Scale to assess Unawareness of Mental Disorder (SUMD) score | Baseline and 3 months after the last tDCS session
  SMUD score (Scale to assess Unawareness of Mental Disorder score) assesses the effect of tDCS on patients' attitudes toward treatment of schizophrenia
Medication Adherence rating Scale (MARS) score | Baseline and 3 months after the last tDCS session
  MARS score assesses the effect of tDCS on patients' attitudes toward treatment of schizophrenia
Brief Medication Questionnaire (BMQ) scores | Baseline and 3 months after the last tDCS session
  BMQ scores (BMQ and BMQ tDCS) assesses the effect of tDCS on patients' attitudes toward treatment of schizophrenia
Source monitoring test score | Baseline and day 5 (after 10-sessions of tDCS regimen)
  Source memory test is performed at baseline and after 10-sessions of tDCS regimen to investigate the effect of tDCS on source monitoring capacities, a cognitive function that may underlie psychotic symptoms (Brunelin et al. 2006).
Functional magnetic resonance imaging (MRI) | Baseline, day 5 (after 10-sessions of tDCS regimen) and 1 month after the last tDCS session
  In order to evaluate treatment-related changes in functional brain connectivity, a functional MRI scans is performed at baseline (day 0), after 10-sessions of tDCS regimen (day 5) and 1 month after the last tDCS session (day 30).
Anatomical magnetic resonance imaging (MRI) | Baseline, day 5 (after 10-sessions of tDCS regimen) and 1 month after the last tDCS session
  In order to evaluate treatment-related changes in functional brain connectivity, an anatomical MRI scans is performed at baseline (day 0), after 10-sessions of tDCS regimen (day 5) and 1 month after the last tDCS session (day 30).
Total serum Brain-Derived-Neurotrophic Factor (BDNF) | Baseline
  Total serum BDNF level is measured to investigate the association between neural markers and clinical response to tDCS. It is hypothised that total serum BDNF is a predictive neural marker of therapeutic response.
Serum Brain-Derived-Neurotrophic Factor (BDNF) isoforms | Baseline
  Serum BDNF isoforms level is measured to investigate the association between neural markers and clinical response to tDCS. It is hypothised that serum BDNFisoforms is a predictive neural marker of therapeutic response.
Self-evaluation of Negative Symptoms (SNS) score | Baseline, 1 month and 3 months after the last tDCS session
  The Self-evaluation of Negative Symptoms scale is a French self-administered questionnaire composed of 20 items organized into 5 domains of negative symptoms of schizophrenia (social withdrawal, diminished emotional range, alogia, avolition, anhedonia).
Fargerström test score | Baseline, 1 month and 6 months after the last tDCS session
  The Fargerström test for nicotine dependence (FTND) is a short form includes six questions designed to estimate the degree of nicotine dependence in tobacco smoking.

CONTACTS AND LOCATIONS:
Locations (10):
- France (9):
  - Centre Hospitalier Le Vinatier - Service de Psychiatrie Adulte, Bron
  - Centre Esquirol - CHU de Caen - Service de Psychiatrie Adulte,, Caen
  - CHU de Clermont-Ferrand - Pôle de Psychiatrie B, Clermont-Ferrand
  - Hôpital Fontan - CHRU de Lille - Pôle de Psychiatrie, Lille
  - Hôpital Edouard Herriot - Service d'Urgences Psychiatriques, Lyon
  - Hôpital de la Colombière - CHU Montpellier - Service de Psychiatrie Adulte, Montpellier
  - Centre Hospitalier Saint-Anne - Service de Psychiatrie Adultes, Paris
  - CHU de St-Etienne - Service d'Urgences Psychiatriques, Saint-Etienne
  - CHRU de Tours - Clinique Psychiatrique Universitaire, Tours
- Centre Hospitalier Princesse Grace - Service de Psychiatrie, Monaco, Monaco

REFERENCES:
- [Result] Brunelin J, Mondino M, Haesebaert J, Attal J, Benoit M, Chupin M, Dollfus S, El-Hage W, Galvao F, Jardri R, Llorca PM, Magaud L, Plaze M, Schott-Pethelaz AM, Suaud-Chagny MF, Szekely D, Fakra E, Poulet E. Examining transcranial random noise stimulation as an add-on treatment for persistent symptoms in schizophrenia (STIM'Zo): a study protocol for a multicentre, double-blind, randomized sham-controlled clinical trial. Trials. 2021 Dec 28;22(1):964. doi: 10.1186/s13063-021-05928-9. PMID 34963486